CLINICAL TRIAL: NCT03609372
Title: Improving HPV Vaccination Delivery in Pediatric Primary Care: The STOP-HPV Trial 6. Single Arm Evaluation of the Maintenance of the STOP-HPV Bundle
Brief Title: The STOP-HPV Trial 6: Single Arm Evaluation of the Maintenance of the STOP-HPV Bundle
Acronym: STOP-HPV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: With the pandemic, we needed to take a 15 month pause in between earlier RCTs. This RCT no longer made sense to conduct.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, Executive Vice-Chair and Vice-Chair for Research, Department of Pediatrics, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6R01CA202261 (NIH); R01CA202261 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-08-01 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Vaccination; Immunization
Keywords: HPV; Vaccination; Practice Based Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): These practices, which previously received the addition of performance feedback and provider prompts in the presence of communication skills training, will receive The STOP-HPV Trial 6: Maintenance
  Interventions: Behavioral: The STOP-HPV Trial 6: Maintenance

INTERVENTIONS:
Behavioral: The STOP-HPV Trial 6: Maintenance — In this period, study team support will be withdrawn after previous bundled intervention (including HPV vaccine communication, performance feedback and provider prompts) was given to reduce MOs and increase HPV vaccination rates.

SUMMARY:
Most adolescents who receive human papillomavirus (HPV) vaccine are vaccinated in pediatric practices, yet missed opportunities (MOs) for HPV vaccination occur often and lead to low HPV vaccination rates. This single arm evaluation (embedded within arm 1 of a 2-arm cluster randomized clinical trial (RCT)) will test the sustainability of improvement made in response to a bundled intervention including HPV vaccine communication, performance feedback and provider prompts to reduce MOs and increase HPV vaccination rates.

DETAILED DESCRIPTION:
HPV vaccine rates remain lower than rates for other adolescent vaccines. Missed opportunities (MOs) are healthcare visits during which a patient is eligible, but does not receive a vaccine. MOs for vaccination contribute strongly to low HPV vaccination rates. This single arm evaluation (embedded within arm 1 of a 2-arm cluster RCT) will test the sustainability of improvement made in repose to a bundled intervention including HPV vaccine communication (done through online educational modules and live office practice sessions), performance feedback reports (that pull from electronic health record (EHR) data, and compare participants performance to their own previous performance and those of others) and provider prompts (via EHR and also office staff prompts, e.g., placing Vaccine Information Statements (VISs) on desk) to reduce MOs and increase HPV vaccination rates.

ELIGIBILITY:
Practice Inclusion Criteria:

* The practice provides HPV vaccination services to adolescents.
* The practice is part of Physician's Computer Company (PCC), Office Practicum (OP) or (a) yet-to-be selected health system(s).
* The practice has had the same EHR system in place for a year or more (with special consideration on a case by case basis if they are close to but not do not reach a year).
* The practice agrees to not participate in other HPV-related QI projects or research interventions during the study period (with special consideration on a case by case basis).

Practice Exclusion Criteria:

* The practice plans to change EHR systems in the next three years.
* The practice participated in the last year, is currently engaged in, or plans to participate in an office-based HPV-related quality improvement (QI) project or research intervention during the study period (with special consideration on a case by case basis).
* Estimated 20% or more of adolescents at the practice receive HPV vaccinations at schools or health department clinics (given standard practice and published data, the investigators expect that few to no practices will need to be excluded based on this restriction).

Patient inclusion criteria:

-All patients of participating practices (intervention and comparison) aged 11-17 years who have at least 1 visit to the practice within the past two years.

Patient exclusion criteria:

-None apart from age of patients (above).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of missed vaccination opportunities among all clinicians | Monthly from months 0 (baseline) through month 27 (end of maintenance period), where month 0 is site specific and depends on completion of site staff training and readiness to proceed.
  Change in the rate of missed vaccination opportunities from baseline through the end of the maintenance period among all clinicians, with a focus on the contrast between the end of the bundled intervention and the maintenance period.
Change in the rate of missed vaccination opportunities among consenting clinicians | Monthly from months 0 (baseline) through month 27 (end of maintenance period), where month 0 is site specific and depends on completion of site staff training and readiness to proceed.
  Change in the rate of missed vaccination opportunities from baseline through the end of the maintenance period among consenting clinicians, with a focus on the contrast between the end of the bundled intervention and the maintenance period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagry, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: No